CLINICAL TRIAL: NCT05045066
Title: MC210501 Differences in Immunological Effects of Vitamin D Replacement Among Black/ African American (AA) Prostate Cancer Patients With Localized Versus Metastatic Disease
Brief Title: Immunological Effects of Vitamin D Replacement Among Black/African American Prostate Cancer Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC210501; HT94252411104 (Other Grant/Funding Number: Department of Defense); PC230672P11 (Other Grant/Funding Number: Department of Defense); NCI-2021-08987 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-004555 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2021-08-25; First posted 2021-09-16 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Localized Prostate Carcinoma; Stage IV Prostate Cancer AJCC v8; Locally Recurrent Prostate Carcinoma; Metastatic Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cholecalciferol; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cholecalciferol) (Experimental): Patients with low vitamin D3 levels receive cholecalciferol PO daily for 8 weeks in the absence of unacceptable toxicity. Patients undergo blood sample collection throughout the study.
  Interventions: Dietary Supplement: Cholecalciferol; Other: Quality-of-Life Assessment; Procedure: Biospecimen Collection

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — Given PO
  Other Names: 9,10-Secocholesta-5,7,10(19)-trien-3-ol; Calciol; Delsterol; Vitamin D3
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
This early phase I is to find out how common vitamin D insufficiency is among African American patients with a history of prostate cancer that has not spread to other parts of the body (localized) or has spread to other places in the body (metastatic) and how vitamin D insufficiency affects the immune system. This study also aims to find out if replacing vitamin D results in normalization of the immune function. Information from this study may benefit prostate cancer patients by identifying vitamin D insufficiency which in several studies had been found to contribute to more aggressive prostate cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the changes in circulating immunological cell function among patients with vitamin D insufficiency and the effects of vitamin D replacement on those changes.

SECONDARY OBJECTIVES:

I. Determine the prevalence of vitamin D insufficiency among black / African American (AA) prostate cancer patients.

II. Determine if there are differences in the peripheral blood immunological cell function in black/AA patients with metastatic or locally recurrent prostate cancer compared to those with localized prostate cancer.

III. Determine if vitamin D replacement is associated with improvement in prostate-specific antigen (PSA) progression free survival (PSA-PFS) of black/AA patients with prostate cancer with detectable changes in immune response compared to those with no detectable changes in immune response and compared to stage matched historical controls.

CORRELATIVE OBJECTIVE:

I. Determine if there are differences in the peripheral blood immunological cell function in Black/AA patients compared to West African/Black patients from Nigeria.

OUTLINE:

Patients with low vitamin D3 levels receive cholecalciferol orally (PO) daily for 8 weeks in the absence of unacceptable toxicity. Patients undergo blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 56 days and then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Pre-Registration:

  * African American males, age >= 18 years
  * Patients with a previous history of localized or metastatic or locally recurrent prostate cancer
* Registration:

  * Patients with Vitamin D levels below 30 ng/ml

Exclusion Criteria:

* Pre-Registration:

  * Known hypersensitivity to vitamin D
  * End stage renal failure on dialysis
  * Liver cirrhosis
  * Currently taking a vitamin D or multivitamin supplement, that has more than 400 IU/10mcg of vitamin D daily for the past month
  * Legal inability or restricted legal ability, medical or psychological conditions not allowing proper study completion or informed consent signature
  * Chemotherapy or surgery or radiation within the last 3 weeks prior to blood collection
  * History of hypercalcemia
* Registration:

  * Chemotherapy or surgery or radiation within the last 3 weeks prior to blood collection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-12-29 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in circulating immunological cell function | Baseline; 8 weeks
  Participants will have blood drawn to measure serum levels of 25-hydroxyvitamin D (25OHD) and to determine immune response. Laboratory endpoints for the levels of antigen-specific T cells and antibodies before and after vitamin D supplementation will be compared. A participant will be considered to have responded if they have developed a ≥3-fold increase in antigen-specific T cells or antibodies at 8 weeks. If T-cell immunity is undetectable, a positive response will be defined as ≥50 antigen-specific T cells/million PBMCs.

SECONDARY OUTCOMES:
Prevalence of vitamin D insufficiency | Baseline; 8 weeks
  Participants will have blood drawn to measure serum levels of 25OHD. The mean and median 25OHD level will be estimated, as well as the percentage of participants that have low vitamin D levels (<30 ng/mL).
Differences in the peripheral blood immunological cell function | Baseline; 8 weeks
  Levels of antigen-specific T cells and antibodies before and after vitamin D supplementation will be compared between black/AA patients with metastatic or locally recurrent prostate cancer and those with localized prostate cancer
Vitamin D replacement association with PSA progression free survival (PSA-PFS) | Up to 3 years
  Participants with detectable changes in immune response will be compared to those with no detectable changes in immune response and compared to stage-matched historical controls to determine whether vitamin D replacement is associated with improvement in PFA-PFS.

OTHER OUTCOMES:
Change in Quality of Life | Baseline; 8 weeks
  Assessed by the Human Services' Centers for Disease Control and Prevention (CDC) Health-Related Quality of Life (HRQOL) Healthy Days Questionnaire. The questionnaire consists of 144 questions about an individual's self-rated general health over the past 30 days. Questions ask about the number of days for which mental and physical health was not good (# of days, none, or don't know/not sure) and whether poor mental or physical health days affected usual activities (yes, no, or don't know/not sure). A higher score (more healthy days) reflects better physical and mental well-being, while a lower score (more unhealthy days) indicates a greater impact from poor physical or mental health and activity limitations.
Difference in peripheral blood immunological cell function by population | Up to 3 years
  A similar parallel study is being conducted at the University of Ilorin in Ilorin, Nigeria. Immunological results from the study at Mayo Clinic will be compared retrospectively with the results from the study in Nigeria under a separate study protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Colon-Otero, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials